CLINICAL TRIAL: NCT03757572
Title: Secondary Intention Wound Healing, in Patients Subjected to Surgical Resection of Pilonidal Cyst, Using Alginate Dressings With Silver and High-G Cellulose, Compared to the Use of Simple Gauze Dressings: Examination of the Quality of Life
Brief Title: Alginate Dressings Versus Gauge Dressings After Pilonidal Cyst Resection: Examination of the Quality of Life
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination due to COVID-19 pandemic. Suspension of elective case operations. Decreased recruitment rate. Inability to reach the estimated sample size.
Sponsor: Larissa University Hospital (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Mamaloudis Ioannis, Principal Investigator, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pilonidal QoL
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Pilonidal Cyst/Fistula
Keywords: Pilonidal; Fistula; Cyst; Alginate; Gauze; Dressings; Prospective; Randomized Controlled Trial
MeSH Terms: conditions — Fistula; Cysts

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding will exist at the level of the investigator who will record the data postoperatively. There will be no blinding at the level of the surgeon or the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alginate dressings (Experimental): The pilonidal cyst will be resected, with the use of a scalpel and then haemostasis will be performed with diathermy.
  Alginate dressings with silver and high-G cellulose, which combine increased absorption properties, antimicrobial action and high coherence will be used. The size of the dressings will be 3cm X 45cm and 1 cm cord will be used for filling the wound cavity. Dressings with perimetric adhesive layer from natural materials for latent breathing of the skin with dressing dimensions based on the wound size, will be also placed.
  Wound care will be performed in a specific way each time that the dressings will be removed. The wound will be irrigated with normal saline and betadine solution and finally without pressure the trauma will be dried.
  Interventions: Other: Alginate dressings
- Simple gauze dressings (Active Comparator): The pilonidal cyst will be resected, with the use of a scalpel and then haemostasis will be performed with diathermy.
  Wound care will be performed with the application of simple gauze dressings. Wound care will be performed in a specific way each time that the dressings will be removed. The wound will be irrigated with normal saline and betadine solution and finally without pressure the trauma will be dried.
  Interventions: Other: Simple gauze dressings

INTERVENTIONS:
Other: Alginate dressings — The pilonidal cyst will be resected, with the use of a scalpel and then haemostasis will be performed with diathermy. Alginate dressings with silver and high-G cellulose will be applied to the wound. The size of the dressings will be 3cm X 45cm and 1 cm cord will be used for filling the wound cavity. Dressings with perimetric adhesive layer from natural materials, will be also placed.
  During wound care the wound will be irrigated with normal saline and betadine solution and finally without pressure the trauma will be dried.
  Arms: Alginate dressings
Other: Simple gauze dressings — The pilonidal cyst will be resected, with the use of a scalpel and then haemostasis will be performed with diathermy. Simple gauze dressings will be applied to the wound.
  During wound care the wound will be irrigated with normal saline and betadine solution and finally without pressure the trauma will be dried.
  Arms: Simple gauze dressings

SUMMARY:
The purpose of this study is to compare the application of alginate dressings with silver and high-G cellulose and the use of simple gauge dressings in patients submitted to surgical resection of pilonidal cyst. The present trial will focus on the postoperative quality of life during the secondary intention wound healing.

DETAILED DESCRIPTION:
Pilonidal cyst was first described by Hodges in 1880. The disease of pilonidal cyst is also known as "Jeep disease", due to the fact that, during World War II (1941-1945), several American soldiers (about 80,000) suffered from this disease, because, either they were driving for long hours on uneven, destroyed by war, roads, or, they were spending time sitting at military vehicles like jeep, trucks and tankers, resulting in being submitted to surgical operation, in order to alleviate the arousing pilonidal cyst problem, at USA military hospitals.

Pilonidal cyst, is considered as one of the most common diseases of the subcutaneous tissues of the sacrococcygeal region. This situation is the result of hair penetrating into the skin, a situation not uncommon in this anatomical area. In a study including 50,000 college students, pilonidal cyst occurrence, in males, was 1.1%, which was 10 times higher compared to females, although a considerable rate of them was asymptomatic. Evidence from studies in England, also, indicate that the disease is more frequent in men than women (1 to 3) . The disease is more common in Caucasians than in Asians or Africans due to the differences in their hair characteristics and the respective hair development pattern. Risk factors include the following: sedentary life (44%), positive family history (38%), obesity (50%) and regional irritation (34%). The disease usually presents during the age of 16 - 20 and prevalence is decreasing drastically after the 25th year of age. This disease rarely develops before the adolescence and after the 40th year of age.

Treatment usually depends on the condition of the disease. An acute abscess is usually controlled with incision and drainage. A chronic pilonidal cyst is best treated with a surgical procedure that involves complete resection of the cyst along with the coexisting fistulas, in order to ensure the minimum reoccurrence rate. There are two choices after surgical resection, secondary intention wound healing or primary trauma closure, with or without a flap. The surgical procedure can be performed with the administration of local anaesthesia in the outpatient office or in a day-clinic, or with the use of general anaesthesia depending on the condition of the patient.

Post operatively secondary intention wound healing is applied in many cases, especially when factors like infection, necrotic tissue or inflammatory tissue are introduced. There are many dressings that can be used for the care of a surgical trauma. The ideal dressing used should have some special characteristics such as absorption of exudates without leakage, provision of a dry environment that prevents bacteria from entering the wound and facilitation of easy appliance, as well as removal. Choosing the right dressing is not based on a certain protocol, but mostly on the surgeon preference.

The current study aims at comparing two groups of patients that will be subjected to surgical resection of pilonidal cyst and secondary intention wound healing. In the first group, dressings like alginate cord with silver and high G cellulose will be used for filling of the wound cavity and a hydro-capillary dressing for sealing and waterproofing the wound. In the other group, simple gauze dressings for the coverage of the wound cavity will be used. Comparison of the two groups will involve all the endpoints that indicate whether such dressings can facilitate faster wound healing, enabling, thus, patients to faster return to their everyday activities. Furthermore, a parameter that has not been, previously, studied, the quality of life after the surgical excision of the pilonidal cyst, by using the SF - 36 and the Quality of life with Chronic Wound questionnaire, will, also, be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Pilonidal cyst
* Age: 18 to 80 years
* American Society of Anesthesiologists (ASA) score: I, II, III, IV
* Disease stage I,II,III and IV

Exclusion Criteria:

* Pilonidal abscess
* Patient age ≥ 80 years or < 18 years
* Pilonidal abscess

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-12-25 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-04-25 (Actual)

PRIMARY OUTCOMES:
Wound healing time | Maximum time frame 50 days postoperatively
  Postoperative required time for wound healing. Measurement unit: days

SECONDARY OUTCOMES:
Postoperative return to everyday activities | Maximum time frame 50 days postoperatively
  Time required for returning to everyday activities. Measurement unit: days
Postoperative pain level | 7, 14, 21, 28, 35, 42 and 49 days postoperatively
  Pain level after surgery, quantified with the use of the Visual Analogue Scale (0-10). Better outcome: 0, Worse outcome: 10. There will be no subscales or total scores.
Postoperative analgesics consumption | 7, 14, 21, 28, 35, 42 and 49 days postoperatively
  Number of analgesic pills consumed per day after surgery. Measurement unit: pills per day
Overall satisfaction level | 50 days postoperatively
  Satisfaction level after surgery, quantified with the use of the Visual Analogue Scale (0-10). Better outcome: 10, Worse outcome: 0. There will be no subscales or total scores.
Cost of the material | Maximum time frame 50 days postoperatively
  Overall cost of the dressings applied
Wound care visits | 7, 14, 21, 28, 35, 42 and 49 days postoperatively
  Number of required visits for postoperative wound care for each patient per week.
Trauma secretions | 7, 14, 21, 28, 35, 42 and 49 days postoperatively
  Trauma secretions leading to extra dressing care. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Wound contamination | Maximum time frame 50 days postoperatively
  Contamination of the wound trauma. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Wound erythema | Maximum time frame 50 days postoperatively
  Erythema of the wound. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Wound haematoma | Maximum time frame 50 days postoperatively
  Haematoma of the wound. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Disease recurrence | Maximum time frame 1 year postoperatively
  Disease recurrence rate. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Difference in the quality of life of the patient | 7, 14 and 21 days potoperatively
  Difference in the quality of life of the patient based on the Quality of Life with Chronic Wounds Wounds (Qol) Questionnaire. 17 items in total. Each item quantified with the use of a Visual Ordinal Scale (0='not at all' to 4='very much'). Global score computed by averaging all items. In total 3 subscales calculated by averaging the respective items:
  Body: Items #1 to #5. Psyche: Items #6 to #10. Everyday life: Items #11 to #16.
Medium term quality of life | 28 days postoperatively
  Quality of life of the patient based on the Short Form 36 (SF-36) questionnaire. 36 items in total. The following ordinal scales will be used for the respective items:
  1 (Better)-5 (Worse): #1, #2, #20, #22, #34, #36.
  1 (Worse)-3 (Better): #3, to #12.
  1 (Worse)-2 (Better): #13, to #19.
  1 (Better)-6 (Worse): #21, #23, #26, #27, #30.
  1 (Worse)-6 (Better): #24, #25, #28, #29, #31.
  1 (Worse)-5 (Better): #32, #33, #35. In total 8 subscales calculated by averaging the respective items. Physical functioning: #3 to #12. Role limitations due to physical health: #13 to #16. Role limitations due to emotional problems: #17 to #19. Energy/fatigue: #23, #27, #29, #31. Emotional well-being: #24 to #26, #28, #30. Social functioning: #20, #32. Pain: #21, #22. General health: #1, #33 to #36.
Treatment satisfaction | 35 days postoperatively
  Patient satisfaction regarding the treatment quantified with the use of a Visual Ordinal Scale (1-5). Better outcome: 5, Worse outcome: 1. There will be no subscales or total scores.
Treatment acceptance | 35 days postoperatively
  Patient acceptance regarding the re-application of the treatment quantified with the use of a Visual Ordinal Scale (1-5). Better outcome: 5, Worse outcome: 1. There will be no subscales or total scores.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Mamaloudis, Principal Investigator — Department of Surgery, University Hospital of Larissa; Konstantinos Tepetes, Study Director — Department of Surgery, University Hospital of Larissa
Locations (1):
- University Hospital of Larissa, Larissa, Greece

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] DWIGHT RW, MALOY JK. Pilonidal sinus; experience with 449 cases. N Engl J Med. 1953 Dec 3;249(23):926-30. doi: 10.1056/NEJM195312032492303. No abstract available. PMID 13111384
- [Background] BUIE LA, CURTISS RK. Pilonidal disease. Surg Clin North Am. 1952 Aug:1247-59. No abstract available. PMID 14950701
- [Background] Berry DP. Pilonidal sinus disease. J Wound Care. 1992 Sep 2;1(3):29-32. doi: 10.12968/jowc.1992.1.3.29. PMID 27911182
- [Background] Sondenaa K, Andersen E, Nesvik I, Soreide JA. Patient characteristics and symptoms in chronic pilonidal sinus disease. Int J Colorectal Dis. 1995;10(1):39-42. doi: 10.1007/BF00337585. PMID 7745322
- [Background] Kronborg O, Christensen K, Zimmermann-Nielsen C. Chronic pilonidal disease: a randomized trial with a complete 3-year follow-up. Br J Surg. 1985 Apr;72(4):303-4. doi: 10.1002/bjs.1800720418. PMID 3886069
- [Background] Sondenaa K, Diab R, Nesvik I, Gullaksen FP, Kristiansen RM, Saebo A, Komer H. Influence of failure of primary wound healing on subsequent recurrence of pilonidal sinus. combined prospective study and randomised controlled trial. Eur J Surg. 2002;168(11):614-8. doi: 10.1080/11024150201680007. PMID 12699097
- [Background] Karydakis GE. New approach to the problem of pilonidal sinus. Lancet. 1973 Dec 22;2(7843):1414-5. doi: 10.1016/s0140-6736(73)92803-1. No abstract available. PMID 4128725
- [Background] Schultz GS, Sibbald RG, Falanga V, Ayello EA, Dowsett C, Harding K, Romanelli M, Stacey MC, Teot L, Vanscheidt W. Wound bed preparation: a systematic approach to wound management. Wound Repair Regen. 2003 Mar;11 Suppl 1:S1-28. doi: 10.1046/j.1524-475x.11.s2.1.x. PMID 12654015
- [Background] Gruessner U, Clemens M, Pahlplatz PV, Sperling P, Witte J, Rosen HR; Septocoll Study Group. Improvement of perineal wound healing by local administration of gentamicin-impregnated collagen fleeces after abdominoperineal excision of rectal cancer. Am J Surg. 2001 Nov;182(5):502-9. doi: 10.1016/s0002-9610(01)00762-0. PMID 11754859
- [Background] Lewis R, Whiting P, ter Riet G, O'Meara S, Glanville J. A rapid and systematic review of the clinical effectiveness and cost-effectiveness of debriding agents in treating surgical wounds healing by secondary intention. Health Technol Assess. 2001;5(14):1-131. doi: 10.3310/hta5140. PMID 11399237
- [Background] Armstrong JH, Barcia PJ. Pilonidal sinus disease. The conservative approach. Arch Surg. 1994 Sep;129(9):914-7; discussion 917-9. doi: 10.1001/archsurg.1994.01420330028006. PMID 8080372
- [Background] Clothier PR, Haywood IR. The natural history of the post anal (pilonidal) sinus. Ann R Coll Surg Engl. 1984 May;66(3):201-3. PMID 6721409
- [Background] Blanco G, Giordano M, Torelli I. [Surgical treatment of pilonidal sinus with open surgical technique]. Minerva Chir. 2003 Apr;58(2):181-7. Italian. PMID 12738928
- [Background] Al-Salamah SM, Hussain MI, Mirza SM. Excision with or without primary closure for pilonidal sinus disease. J Pak Med Assoc. 2007 Aug;57(8):388-91. PMID 17902520
- [Background] Irkorucu O, Erdem H, Reyhan E. The best therapy for pilonidal disease: which management for which type? World J Surg. 2012 Mar;36(3):691-2. doi: 10.1007/s00268-011-1285-2. No abstract available. PMID 21956594
- [Background] Anagnostopoulos F, Niakas D, Pappa E. Construct validation of the Greek SF-36 Health Survey. Qual Life Res. 2005 Oct;14(8):1959-65. doi: 10.1007/s11136-005-3866-8. PMID 16155784
- [Background] Blome C, Baade K, Debus ES, Price P, Augustin M. The "Wound-QoL": a short questionnaire measuring quality of life in patients with chronic wounds based on three established disease-specific instruments. Wound Repair Regen. 2014 Jul-Aug;22(4):504-14. doi: 10.1111/wrr.12193. PMID 24899053
- [Background] Deutsch CJ, Edwards DM, Myers S. Wound dressings. Br J Hosp Med (Lond). 2017 Jul 2;78(7):C103-C109. doi: 10.12968/hmed.2017.78.7.C103. No abstract available. PMID 28692373

DOCUMENTS (2):
  • Study Protocol (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03757572/Prot_000.pdf
  • Informed Consent Form (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03757572/ICF_001.pdf